CLINICAL TRIAL: NCT07110090
Title: A Dose-Escalation Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Umbilical Cord Blood Megakaryocyte Injection (XJ-MK-002) in Patients With Cancer Therapy-Induced Thrombocytopenia (CTIT)
Brief Title: Umbilical Cord Blood Megakaryocyte Injection (XJ-MK-002) for Cancer Therapy-Induced Thrombocytopenia (CTIT)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM_XJ-MK-002
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Thrombocytopenia; Cancer
MeSH Terms: conditions — Thrombocytopenia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose level (Experimental): 1.0×108 cells per person.
  Interventions: Biological: Umbilical Cord Blood Megakaryocyte Injection (XJ-MK-002)
- medium dose level (Experimental): 3.0×108 cells per person
  Interventions: Biological: Umbilical Cord Blood Megakaryocyte Injection (XJ-MK-002)
- high dose level (Experimental): 6.0×108 cells per person
  Interventions: Biological: Umbilical Cord Blood Megakaryocyte Injection (XJ-MK-002)

INTERVENTIONS:
Biological: Umbilical Cord Blood Megakaryocyte Injection (XJ-MK-002) — dosage form: Injection dosage: 10 mL/bag, 1×10⁷ cells/mL frequency: Each subject will be administered a single infusion of XJ-MK-001 at their respective enrolled dose level.

SUMMARY:
This study is a single-center, open-label, single-arm, dose-escalation clinical trial to assess safety & tolerability of XJ-MK-002 in CTIT patients. It plans to recruit subjects aged 18 to 75 years old with chemotherapy-induced thrombocytopenia (CTIT). The study is designed with three dose levels: low dose (1.0×108 viable cells per person), medium dose (3.0×108 viable cells per person), and high dose (6.0×108 viable cells per person). The first dose group (low dose) will enroll one subject for accelerated titration, while the other two dose groups will enroll at least three subjects each. Subjects successfully enrolled will receive only one cell therapy session. After the cell therapy, they will undergo a 28-day dose-limiting toxicity (DLT) observation period.

DETAILED DESCRIPTION:
XJ-MK-002 injection is a cord blood-derived megakaryocyte suspension, which, following intravenous infusion, undergoes differentiation and fragmentation into platelets under hemodynamic shear stress and physiological regulation within the in vivo environment, thereby elevating platelet levels. The primary endpoint of this study is:

• Incidence and severity of adverse events within 28 days.

Secondary endpoints include:

* Incidence and severity of adverse events during the trial period;
* Evaluation of changes in platelet counts from baseline at 1h, 2h, 4h, D2, D3, D7, D14, and D28 after XJ-MK-002 infusion.

Exploratory endpoints comprise:

* Assessment of the modified platelet recovery rate (PPR) and corrected count increment (CCI) at 1h, 2h, 4h, D2, D3, D7, D14, and D28 post-infusion of XJ-MK-002;
* Investigation of the pharmacokinetic parameters of XJ-MK-002, including but not limited to Cmax, Tmax, and AUC0-t.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 75 years (inclusive) at the time of signing the informed consent, regardless of gender.
2. Histologically and/or cytologically confirmed diagnosis of a malignant tumor, with thrombocytopenia due to anti-tumor treatments (e.g., chemotherapy, immunotherapy, targeted therapy, and radiotherapy), 50×10⁹/L≤platelet count (PLT) is ≤100×10⁹/L, confirmed by blood tests (with reconfirmation on the day prior to infusion) and with no bleeding
3. No transfusion of platelets or blood products containing platelet components within 72 hours prior to investigational product administration.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
5. Estimated life expectancy of more than 3 months.
6. Female subjects of childbearing potential (WOCBP) and male subjects with WOCBP partners must agree to use highly effective contraception methods in accordance with ICH M3 (R2) guidelines during the trial and for 6 months after administration. Male subjects must also agree not to donate sperm during this period. WOCBP must have a negative pregnancy test result within 7 days prior to enrollment.

Exclusion Criteria:

1. History of platelet transfusion refractoriness.
2. History of severe allergic reactions related to blood transfusion.
3. History of bleeding disorders or thrombocytopenia caused by conditions other than CTIT.
4. Splenomegaly or hypersplenism.
5. Use of thrombopoietin-stimulating drugs within 7 days prior to receiving the investigational product, including recombinant human thrombopoietin (rhTPO), recombinant human interleukin-11 (rhIL-11), romiplostim, eltrombopag, hetrombopag, leucogen tablets, aminopeptidase tablets, and caffeic acid tablets.
6. Subjects with existing severe bleeding (e.g., cerebral hemorrhage, severe gastrointestinal bleeding, or severe hemoptysis).
7. Subjects with hemophilia or coagulation disorders.
8. History of thromboembolic diseases (deep vein thrombosis, arterial thrombosis) within 6 months before screening, or patients with catheter-related thrombosis within 1 month before screening.
9. History of cardiac diseases within 3 months before screening, or a history of severe cardiovascular diseases (e.g., congestive heart failure (NYHA Class 3/4), known arrhythmias that increase the risk of thromboembolic events (e.g., atrial fibrillation, atrial flutter, unstable angina), coronary stent placement, angioplasty, or coronary artery bypass grafting).
10. Major organ surgery (excluding needle biopsy) or severe trauma within 4 weeks before administration of the investigational product or anticipated major surgery during the trial.
11. Use of anticoagulant drugs within 7 days before screening, including vitamin K antagonists, low molecular weight heparin (except for minimal heparin use for catheter locking), factor Xa inhibitors (e.g., rivaroxaban), thrombin inhibitors, and/or antiplatelet therapy (e.g., aspirin).
12. Coagulation function abnormalities: activated partial thromboplastin time (APTT) >1.5× upper limit of normal (ULN); international normalized ratio (INR) >1.5×ULN.
13. Liver and kidney function abnormalities: liver function (for non-liver cancer patients or those without liver metastasis): total bilirubin (TBIL) >2.5×ULN, alanine aminotransferase (ALT) >2.5×ULN, aspartate aminotransferase (AST) >2.5×ULN; renal function: creatinine clearance (Ccr) <50 mL/min, or serum creatinine (Cr) >1.5×ULN.
14. Complete blood count abnormalities: Absolute neutrophils count <1.0×109/L, hemoglobin <80g/L (use of erythropoietin infusion therapy according to clinical standards is allowed during screening).
15. Positive serology tests during screening: positive anti-HIV antibody or anti-treponema pallidum specific antibody test; or positive hepatitis C antibody with HCV RNA copy number above the upper limit of normal, positive hepatitis B surface antigen, or history of hepatitis B infection; or positive hepatitis B core antibody with HBV-DNA ≥2000 IU/mL within the last 3 months before screening.
16. Uncontrolled severe chronic or active infection requiring intravenous antibiotic treatment before administration.
17. Subjects with known allergies to the investigational product, its active ingredients, or any of its excipients.
18. Use of any investigational product with a similar mechanism of action within 4 weeks prior to administration of the investigational product, or current participation in another clinical trial (except for observational, non-interventional clinical trials, or the follow-up period of an interventional clinical trial).
19. History of hematopoietic stem cell transplantation with acute graft-versus-host disease requiring therapeutic intervention.
20. Pregnant or lactating female subjects.
21. Any other medical condition that, in the investigator's judgment, precludes participation in this study or completion of follow-up observations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and relationship to XJ-MK-001 of adverse events within 28 days post-infusion of XJ-MK-002. | within 28 days post-infusion of XJ-MK-002
  Incidence and severity of adverse events within 28 days.

SECONDARY OUTCOMES:
a) The incidence, severity of adverse events and their correlation with XJ-MK-002 during study period. b) Change in platelet counts from baseline to D28 after XJ-MK-002 infusion. | within 180 days post-infusion of XJ-MK-001
  Adverse events were evaluated according to CTCAE 5.0, platelet counts measured by blood routine test.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, Study Director — Clinical Trial Center, National Cancer Center of China
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences 17 Panjiayuan Nanli, Chaoyang District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No